CLINICAL TRIAL: NCT06955741
Title: A Phase 1, Randomized, Open-label, Parallel, Single-dose Study to Assess the Pharmacokinetics, Tolerability, and Absolute Bioavailability of Subcutaneous Administration of BMS-986446, an Anti-MTBR Tau Monoclonal Antibody, in Healthy Participants
Brief Title: A Study to Assess Drug Levels, Tolerability and Absolute Biological Availability of Single-dose of BMS-986446 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN008-0026
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer
Keywords: Bioavailability Study; Subcutaneous Injection; Anti-MTBR Tau Monoclonal Antibody
MeSH Terms: interventions — Acetaminophen; Loratadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: BMS-986446 IV; Drug: Acetaminophen; Drug: Loratadine
- Arm B (Experimental)
  Interventions: Drug: BMS-986446 SC; Drug: Acetaminophen; Drug: Loratadine

INTERVENTIONS:
Drug: BMS-986446 IV — Specified dose on specified days was administered intravenously (IV).
  Arms: Arm A
Drug: BMS-986446 SC — Specified dose on specified days was administered subcutaneously (SC).
  Arms: Arm B
Drug: Acetaminophen — Specified dose on specified days
Drug: Loratadine — Specified dose on specified days

SUMMARY:
The purpose of this study is to assess drug levels, tolerability and absolute biological availability of single subcutaneous dose of BMS-986446 in healthy participants

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a Body Mass Index (BMI) of 18.0 to 30.0 kg/m2.
* Participants must be healthy as determined by medical history, physical examination, neurological examination, vital signs, 12-lead ECG, C-SSRS, and clinical laboratory evaluations.

Exclusion Criteria:

* Participants must not have clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardiovascular, endocrinological, immune-mediated disorder, hematological, ongoing allergic disorder requiring treatment, metabolic disorder, cancer, or cirrhosis.
* Participants must not have prior exposure to BMS-986446 (PRX005).
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Ratio (GMR) of Maximum Observed Serum Concentration (Cmax) of BMS-986446 Administered IV versus SC | Up to approximately Day 85
GMR of Area Under the Serum Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC(0-T)) of BMS-986446 Administered IV versus SC | Up to approximately Day 85
GMR of Area Under the Serum Concentration-time Curve From Time Zero to 672 Hours (AUC(0-672)) of BMS-986446 Administered IV versus SC | Up to approximately Day 85
Absolute Bioavailability (F) Estimated From GMR of AUC(INF) of BMS-986446 Administered as SC versus IV Infusion | Up to approximately Day 85

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to approximately Day 85
Number of Participants With Serious Adverse Events (SAEs) | Up to approximately Day 85
Number of Participants With AEs Reported Related to BMS-986446 | Up to approximately Day 85
Number of Participants With Clinically Significant Vital Sign Abnormalities | Up to approximately Day 85
Number of Participants With Clinically Significant Changes in 12-lead Electrocardiogram (ECG) | Up to approximately Day 85
Number of Participants With Clinically Significant Physical Examination (PE) Abnormalities | Up to approximately Day 85
Number of Participants With Suicidality as Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to approximately Day 85
Number of Participants With Clinically Significant Laboratory Assessment Abnormalities | Up to approximately Day 85
Cmax of BMS-986446 | Up to approximately Day 85
AUC(0-T) of BMS-986446 | Up to approximately Day 85
AUC(0-672) of BMS-986446 | Up to approximately Day 85
Area Under the Serum Concentration-time Curve From Time Zero Extrapolated to Infinite Time (AUC(INF)) of BMS-986446 | Up to approximately Day 85
Time of Maximum Observed Serum Concentration (Tmax) of BMS-986446 | Up to approximately Day 85
Apparent Terminal Serum Half-life (T-HALF) of BMS-986446 | Up to approximately Day 85
Total Body Clearance in IV Infusion (CLT) of BMS-986446 | Up to approximately Day 85
Apparent Total Body Clearance in SC Administration (CLT/F) of BMS-986446 | Up to approximately Day 85
Volume of Distribution of Terminal Phase in IV Infusion (Vz) of BMS-986446 | Up to approximately Day 85
Apparent Volume of Distribution of Terminal Phase in SC Administration (Vz/F) of BMS-986446 | Up to approximately Day 85
Number of Participants With Anti-drug Antibody Development | Up to approximately Day 85
Local Tolerance Evaluation SC Administration of BMS-986646 Assessed by Questionnaire | Up to approximately Day 85
  Participant-reported response will be obtained using questionnaires that assess for pain (using a Numeric Rating Scale), itching, burning, pressure, and soreness/tenderness at the site injection.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Local Institution - 0001, Anaheim, California
  - Local Institution - 10000, Anaheim, California

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.htm
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com